CLINICAL TRIAL: NCT06956807
Title: First in Human Open Label Multicentre Clinical Trial to Evaluate the Safety and Efficacy of Epicardial Implantation of Collagen Membranes With Allogeneic Adipose Derived Stem Cells in Patients With Ischaemic Left Ventricular Dysfunction Scheduled to Undergo Coronary Revascularisation Surgery
Brief Title: Safety and Efficacy of Epicardial Implantation of Collagen Membranes With Allogeneic Adipose Derived Stem Cells
Acronym: CARDIOMESH II
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Viscofan (Industry)
Collaborators: KCRI Sp. z o.o. (Unknown); Medical University of Silesia (Other); Clinica Universidad de Navarra, Universidad de Navarra (Other); Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARDIOMESH II; 2024-517738-16-00 (EU CTIS Number); 2022-002180-29 (EudraCT Number)
Record Dates: First submitted 2025-04-15; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: CABG-patients; Heart Failure; Myocardial Infarction (MI)
Keywords: heart failure; coronary revascularisation surgery; adipose-derived stem cells; myocardial infarction
MeSH Terms: conditions — Heart Failure; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with VB-C01 (Experimental): Treatment arm in which patients will be treated with a VB-C01 cellularised patch.
  Interventions: Combination Product: VB-C01 cellularised patch

INTERVENTIONS:
Combination Product: VB-C01 cellularised patch — surgical epicardial implantation of a membrane seeded with allogeneic adipose tissue derived stem cells in patients scheduled to undergo coronary revascularisation surgery and at high risk of developing heart failure

SUMMARY:
* The Cardiomesh II clinical trial is a phase I open label study intended to enrol 10 patients to evaluate the safety and efficacy of surgical epicardial implantation of a membrane seeded with allogeneic adipose tissue derived stem cells in patients scheduled to undergo coronary revascularisation surgery and at high risk of developing heart failure.
* The primary objective of the study is to evaluate the safety of surgical implantation of this membrane in patients with large ischaemic myocardial scars scheduled to undergo coronary revascularisation surgery. The secondary objective is to investigate the efficacy of the above treatment in terms of reduction of scar size and ventricular function parameters.

DETAILED DESCRIPTION:
* The clinical trial CARDIOMESH II aims to attenuate adverse remodelling of the left ventricle, which is the main cause of death in ischaemic heart disease, through the development of a new regenerative therapy consisting of the combination of allogeneic adipose derived stem cells with bovine derived collagen membranes to promote repair of damaged myocardium. This is predicted to achieve a 10% reduction in mortality related to ischaemic heart failure.
* Specifically, the working hypotheses of the project are:
* Surgical implantation of a membrane containing allogeneic adipose derived stem cells in patients with large myocardial scars scheduled to undergo coronary revascularisation surgery is technically feasible.
* Surgical implantation of a membrane containing allogeneic adipose derived stem cells in patients with large myocardial scars scheduled to undergo coronary revascularisation surgery is safe in terms of the primary objective consisting of major adverse cardiac and cerebrovascular events (MACCEs).
* Surgical implantation of the aforementioned bioengineering product is safe in terms of cardiac effects and immunological analysis.
* Surgical implantation of this cellularised membrane shows beneficial effects in terms of efficacy measured by surrogate cardiac imaging parameters.
* Designed as an international phase I clinical trial to be conducted at two sites in two European countries, the purpose of the study is to establish the basic safety parameters and to obtain preliminary efficacy data on clearly established surrogate variables to undertake future larger scale trials focused on clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients planning to undergo coronary revascularisation surgery within one month of study entry.
2. LVEF ≤45% by CMRI.
3. History of myocardial infarction at least 3 months prior to inclusion.
4. Scar covering at least 15% of the total left ventricular myocardial mass defined by late enhancement on CMRI.

Exclusion Criteria:

1. Participation in another clinical trial within 30 days prior to inclusion.
2. Prior treatment with cell or gene therapy.
3. Be a candidate for heart transplant at the time of study entry.
4. Diagnosis of acute myocardial infarction with 3 months prior to inclusion.
5. Need for urgent revascularisation surgery.
6. Strict contraindication for the use of CMRI (pacemaker or implantable automatic defibrillator carriers, previous reactions to gadolinium contrast, claustrophobia, cochlear implants, etc.).
7. Presence of uncontrolled ventricular arrhythmias (ventricular tachycardia or ventricular fibrillation) at the time of implant surgery.
8. Active systemic infection.
9. Women who are pregnant or breastfeeding.
10. Mental disease or psychological condition that impedes the subject from understanding the nature of the protocol and granting his/her consent
11. Advanced dementia according to the Barthel index.
12. History of primary or acquired immunodeficiency or on immunosuppressive therapy (within 3 months prior to inclusion or if the need for immunotherapy is foreseeable at any time during the study follow up).
13. Tumour disease, except that eradicated at least 5 years prior to inclusion in the study and without receiving chest radiotherapy. Completely eradicated non melanoma skin tumours (at any time) not requiring chest chemotherapy or radiotherapy are permitted.
14. History of autoimmune disease.
15. Stroke within 12 months prior to inclusion.
16. Respiratory compromise or need for home oxygen therapy.
17. Life expectancy of less than 1 year for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
combination of MACCEs at all follow up visits during the first year after treatment | 12 months
  combination of MACCEs at all follow up visits during the first year after treatment (after surgery, at 1, 3, 6, 9 and 12 months). MACCEs are defined as all cause death, myocardial infarction requiring target vessel revascularisation, hospitalisation for heart failure, cardiac tamponade or pericardial constriction, sustained ventricular tachycardia, ventricular fibrillation, and stroke.

SECONDARY OUTCOMES:
Safety - Composite MACCE | 12 months
  Composite MACCE (all cause death, myocardial infarction requiring target vessel revascularisation, hospitalisation for heart failure, cardiac tamponade or pericardial constriction, sustained ventricular tachycardia, ventricular fibrillation, and stroke) at all follow up visits during the first year after treatment (after surgery, 1, 3, 6, 9 and 12 months),
Safety - Hematology parameters | 12 months
  Erythrocytes, Haemoglobin, Haematocrit, Leukocytes, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils, Platelets, Prothrombin time, APTT, INR.
  Measurement of the values and evaluation of their clinical significance in case they are outside of the normal range.
Safety - Adverse Events | 12 months
  Any cause adverse event at all follow up visits during the first year after treatment (after surgery, 1, 3, 6, 9 and 12 months)
Safety - Biochemical blood parameters | 12 months
  Measurement of biochemistry paramenters in blood including Glucose, Creatinine, Urea, GOT, GPT, GGT, Total bilirubin, Alkaline phosphatase, Total cholesterol, LDL-cholesterol, HDL-cholesterol, Triglycerides, Total proteins, Sodium, Potassium, Calcium, Chloride.
  Evaluation of clinical significance in case values are out of normal range.
Safety - New York Heart Association (NYHA) functional class | 12 months
  Assessment of the New York Heart Association (NYHA) functional class before surgery (the first assessment will be done during the screening process and repeated before the procedure), at 6 and 12 months after surgery.
Safety - Minnesota Living with Heart Failure (MLHFQ) questionnaire | 12 months
  Minnesota Living with Heart Failure (MLHFQ) questionnaire, before surgery (the first assessment will be done during the screening process, at least one day before surgery), at 6 and 12 months after surgery.
Safety - 6 minute walk test | 12 months
  The 6 minute walk test will be performed before surgery (the first assessment will be done during the screening process, at least one day before surgery), at 6 and 12 months after surgery.
Safety - Brain natriuretic peptide curve (Nt proBNP or BNP) | 12 months
  Brain natriuretic peptide curve (Nt proBNP or BNP, depending on the availability at each site using the same parameter throughout the follow up of each patient). Levels will be measured during the screening process (the first assessment will be done, at least one day before surgery), on the second day after surgery and at 6 and 12 months after product administration.
Safety - C reactive protein (CRP) levels | 1 month
  C reactive protein (CRP) levels will be assessed prior to surgery (the first assessment will be done during the screening process, repeated prior to surgery), at hospital discharge, and 1 month after product administration.
Safety - Incidence of subacute pericardial inflammation or constrictive physiology | 12 months
  Incidence of subacute pericardial inflammation or constrictive physiology as assessed by echocardiography and cardiac magnetic resonance imaging (CMRI) at months 1, 6 and 12 after treatment. The first assessment will be done during the screening process.
Safety - Immunological analysis | 1 month
  The following immunological analysis will be performed: B Lymphocytes, NK Lymphocytes (CD16+), T Lymphocytes (CD3+), Th Lymphocytes (CD4+), Activated Th Lymphocytes (CD4+DR+), Treg Lymphocytes (CD4+CD25+), Treg Lymphocytes (CD4+CD25+), Activated Treg Lymphocytes (CD4+CD25+DR+), Cytotoxic T Lymphocytes (CD8+), Activated Cytotoxic T Lymphocytes (CD8+DR+), Cytotoxic Treg Lymphocytes (CD8+CD25+), Activated Cytotoxic Treg Lymphocytes (CD8+CD25+DR+), Albumin, Alpha globulin, Beta globulin, Gamma globulin, IgG, IgM and anti-HLA antibodies (the first assessment will be done during the screening process) at discharge (at discharge excluding Serum Cytokines and anti-HLA antibodies) and 1 month after product administration.
Efficacy - Change in scar size | 12 months
  Absolute change in scar size expressed as percentage of left ventricular mass (i.e. scar mass corrected for total left ventricular mass), absolute change in percentage of viable left ventricular mass (i.e. viable mass corrected for total left ventricular mass), absolute change in total scar size (expressed in grams), and absolute change in viable mass (expressed in grams).
Efficacy - end systolic volume | 12 months
  Biomechanical parameters of the left ventricle: end systolic volume, end diastolic volume, ejection fraction, segmental contractility, and segmental wall thickness. All values will be obtained by CMRI analysis.
Efficacy - end diastolic volume | 12 months
  Biomechanical parameters of the left ventricle: end systolic volume, end diastolic volume, ejection fraction, segmental contractility, and segmental wall thickness. All values will be obtained by CMRI analysis.
Efficacy - ejection fraction | 12 months
  Biomechanical parameters of the left ventricle: end systolic volume, end diastolic volume, ejection fraction, segmental contractility, and segmental wall thickness. All values will be obtained by CMRI analysis.
Efficacy - segmental contractility | 12 months
  Biomechanical parameters of the left ventricle: end systolic volume, end diastolic volume, ejection fraction, segmental contractility, and segmental wall thickness. All values will be obtained by CMRI analysis.
Efficacy - segmental wall thickness | 12 months
  Biomechanical parameters of the left ventricle: end systolic volume, end diastolic volume, ejection fraction, segmental contractility, and segmental wall thickness. All values will be obtained by CMRI analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Radoslaw Gocol, MD, Study Chair — Medical University of Silesia; Javier Bermejo, MD, Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (1):
- Górnośląskie Centrum Medyczne im. prof. Leszka Gieca Śląskiego Uniwersytetu Medycznego w Katowicach, Katowice - Ochojec, Poland

IPD SHARING:
Plan to Share IPD: Undecided